CLINICAL TRIAL: NCT04200196
Title: Improvement of Anxiety Management During a Venous Puncture About Children 3 to 6 Years, with a Participatory Entertainment Method
Brief Title: Improvement of Anxiety Management During a Venous Puncture About Children with a Participatory Entertainment Method
Acronym: PEDIPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC19.0189
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorders
Keywords: anxiety; children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is an interventional prospective controlled study with 2 arms:
  * the "fabrique à histoire" arm : production and listening a story by the children
  * the controlled arm: usual care (to sing, blow up a baloon, etc)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Fabrique à histoire" (Experimental): Children 3 to 6 years in pediatric emergency needing to venous puncture and randomized in the "fabrique à histoire (Lunii(R))" arm in addition to the routine anaesthetic cream patch.
  Interventions: Procedure: "fabrique à histoire"
- Usual care (Active Comparator): Children 3 to 6 years in pediatric emergency needing to venous puncture and randomized in the habitual care arm in addition to the routine anaesthetic cream patch.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: "fabrique à histoire" — "Fabrique à histoire" is a participatory entertainment method. Children of this arm going to create and listening a story before and during the venous puncture.
  Arms: "Fabrique à histoire"
Procedure: Usual care — It is a passive entertainment method. Children of this arm going to do habitual activities before and during the venous puncture, like to sing, blow up a balloon, to play with recreational thing, etc.
  Arms: Usual care

SUMMARY:
The purpose of this study is to demonstrate an anxiety decrease about children 3 to 6 years during a venous puncture with the "fabrique à histoire".

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate an anxiety decrease about children 3 to 6 years during a venous puncture with the "fabrique à histoire".

the study will compare the "fabrique à histoire"(Lunii(R)) with the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 to 6 years in pediatric emergency needing to venous puncture
* Oral consent by children
* Informed and signed consent by tenured of parent authority
* To have Anaesthetic patch 45 minutes or more before the venous puncture

Exclusion Criteria:

* To have Anaesthetic patch less than 45 minutes before the venous puncture because of necessity to blood test or an other emergency
* Necessity to analgesic 3 emergency
* Necessity to MEOPA
* Minor parents
* Assessment of anxiety is not possible because of comorbidity
* Anterior participation to these study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale (mYPAS) | During venipuncture, an average of 1,5 hours
  Evolution of mYPAS (validated anxiety scale with a scale 23,3 (no anxiety) to 100 (max of anxiety) between T0 (before venipuncture) and T1 (venipuncture). mYPAS is quoted by an extern observator
modified Yale Preoperative Anxiety Scale (mYPAS) | through study completion, an average of 2 hours
  Evolution of mYPAS (validated anxiety scale with a scale 23,3 (no anxiety) to 100 (max of anxiety) between T0 and T2 (after venipuncture). mYPAS is quoted by an extern observator.

SECONDARY OUTCOMES:
Children face scale | through study completion, an average of 2 hours
  Evolution of Self-assessment of pain with the face scale caused by the venous puncture for children 4 to 6 years between T0 and T2 (after venipuncture)
FLACC Scale | through study completion, an average of 2 hours
  Evolution assessment of pain caused by the venous puncture for children assess by caregivers and measured with FLACC Scale (Face Legs Activity Cry Consolability / 0=no pain and 10=max pain) between T0 and T2 (after venipuncture)
Parent anxiety assessment | through study completion, an average of 2 hours
  Assessment of anxiety caused by the venous puncture for children assess by parents at T2 with an Analogue and Visual Scale (AVS) 10 levels (0=No anxiety 10=max anxiety)
Parent pain assessment | through study completion, an average of 2 hours
  Assessment of pain caused by the venous puncture for children assess by parents at T2 with an AVS 10 level (0=No pain 10=max pain)
Number of venous puncture before success | through study completion, an average of 2 hours
  Number of venous puncture tentative(s) before success
Venous puncture success | through study completion, an average of 2 hours
  Success or not (Yes/No) of the venous puncture
Time before venous puncture success | through study completion, an average of 2 hours
  Measure of time spent performing the act before its success
Caregivers feedback | through study completion, an average of 2 hours
  Assessment of caregivers feedback from the gesture with an AVS 0 (worst feeling) to 10 (best feeling)
Parents feedback | through study completion, an average of 2 hours
  Assessment of parents feedback from the gesture with an AVS 0 (worst feeling) to 10 (best feeling)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.